CLINICAL TRIAL: NCT00618956
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of Milnacipran 100 And 200 MG Daily in Patients With Fibromyalgia: Effects On 24 Hour Ambulatory Blood Pressure
Brief Title: A Study Of Milnacipran In Patients With Fibromyalgia: Effects On 24 Hour Ambulatory Blood Pressure Monitoring
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Cypress Bioscience, Inc. (Industry)
Responsible Party: Allan Spera, Director, Forest Laboratories, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN-MD-12
Record Dates: First submitted 2008-01-31; First posted 2008-02-20 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Fibromyalgia
Keywords: NSRI; milnacipran; fibromyalgia; blood pressure; hypertension
MeSH Terms: conditions — Fibromyalgia; Hypertension | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Milnacipran hydrochloride
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran hydrochloride — Milnacipran 100 to 200 mg/day tablet (administered in divided doses, twice daily [BID]), oral administration.
  Other Names: Ixel (outside of United States)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
The study is designed to accurately assess any changes in blood pressure and pulse at 100 and 200 mg daily dose of milnacipran in patients with fibromyalgia syndrome.

DETAILED DESCRIPTION:
This study is double blind (neither you nor the physician will know if you are receiving active study drug or placebo, an inactive compound such as a sugar pill) and it is being conducted at various research centers in the United States.

If the study staff determines that you are eligible and you decide to participate, there will be approximately 11 study visits in about 3 months. During these visits, you will undergo routine health exams and complete different kinds of questionnaires.

This study requires that you wear a blood pressure cuff continuously for 24 hours on three separate occasions. You will also be required to make multiple same-day visits to the study site on three separate occasions for blood draws.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in the study, patients must meet the following criteria:

  1. Patients may be male or female between the ages of 18 and 70 years, inclusive
  2. Patients must have been diagnosed of primary fibromyalgia, as defined by the 1990 ACR Criteria for the Classification of Fibromyalgia
  3. Females must be either postmenopausal (no menses for at least 1 year), posthysterectomy, postoophorectomy (bilateral), or, if of childbearing potential, must have a negative urine pregnancy test prior to randomization and be using a medically acceptable form of contraception (eg, hormonal birth control, IUD, double-barrier method [eg, simultaneous use of two of the following: male condom, female condom, diaphragm], or a barrier method plus a spermicidal agent [contraceptive foam, jelly, or cream])
  4. Patients must have the ability to give written informed consent
  5. Patients may have hypertension untreated or treated with a maximum of two antihypertensive medications. (Note: medications contributing to a combination product(s) will each be considered as a separate medication.) If untreated, the patient should be stable, with no expectation of initiating treatment during the study. If treated, the patient must have been on stable doses of antihypertensive medications for at least 2 months, with the expectation that dose adjustments will not be necessary for the duration of the study. A patient will be classified as hypertensive if the patient is taking antihypertensive medication, has a SBP equal to or greater than 130 mm Hg, or has a DBP equal to or greater than 85 mm Hg. A patient will be classified as normotensive if he/she is not on antihypertensive medication and has a SBP less than 130 mm Hg and DBP less than 85 mm Hg
  6. Patients must have a mean of two sitting SBP measurements of less than 160 mm Hg and sitting DBP less than 100 mm Hg at Visit 1 (Screening) and Visit 2 (Baseline/Randomization) using an automatic office blood pressure monitor
  7. Patients must have normal physical examination findings, clinical laboratory results, and electrocardiogram (ECG) results from Visit 1 (Screening) or abnormal findings judged not clinically significant by the Investigator and documented as such in the eCRF
  8. Patients must be willing to withdraw from CNS-active therapies marketed as antidepressants, including monoamine oxidase inhibitors, tricyclics, tetracyclics, selective-serotonin reuptake inhibitors (SSRIs), noradrenaline reuptake inhibitors (NARIs), noradrenaline-serotonin reuptake inhibitors (NSRI), serotonin-noradrenaline reuptake inhibitors (SNRIs), and St. John's Wort
  9. Patients must be willing to withdraw from pregabalin (Lyrica) or gabapentin (Neurontin).
  10. Patients must be willing to withdraw from stimulant medications such as those used to treat attention deficit disorder/attention deficit hyperactivity disorder (eg, amphetamine/dextroamphetamine [Adderall], methylphenidate, dextroamphetamine) or the fatigue associated with sleep apnea or shift work (eg, modafinil)
  11. Patients must be willing to withdraw from anorectic agents such as diethylpropion , sibutramine (Meridia), and phentermine (Adipex)
  12. Patients must be willing to withhold certain medications for the 24 hours before, as well as during, any ABPM assessment. These medications include phosphodiesterase type 5 inhibitors (eg, Viagra, Levitra, Cialis, Edex, Muse), decongestants (eg, pseudoephedrine, phenylephrine), and antimigraine therapies (eg, triptans such as Imitrex and Maxalt, ergotamines such as Cafergot and Midrin). If, for any reason, the patient takes any of these medications, the ABPM visit should be rescheduled so that at least 24 hours have transpired since the patient's last use

Exclusion Criteria:

* Patients who meet any of the following criteria will not be eligible to participate in the study:
* Psychological/Psychiatric Criteria

  1. Patients with a significant risk of suicide, according to the Investigator's judgment or based on an answer of 2 or 3 for question 9 of the Beck Depression Inventory (BDI) (regarding suicidal ideation) performed at Visit 1 (Screening) or Visit 2 (Baseline/Randomization)
  2. Patients with a total BDI score greater than 25 at Visit 1 (Screening) or Visit 2 (Baseline/Randomization)
  3. Patients testing positive for illegal substances prior to Visit 2 (Baseline/Randomization) as demonstrated by positive drug screening or based on the Investigator's judgment
  4. Patients with any history or behavior that would, in the Investigator's judgment, prohibit compliance for the duration of the study
* Somatic Criteria

  1. Patients with myocardial infarction and/or stroke within the past 12 months; active cardiac disease (American Heart Association Functional Class 2, 3, or 4); congestive heart failure; hemodynamically significant valvular heart disease (including patients with a prosthetic heart valve); hypertensive cardiovascular disease changes (heart, eyes or kidneys) that in the Investigator's judgment, would preclude patient participation; ischemic changes; and/or clinically significant cardiac rhythm or conduction abnormalities (including atrial fibrillation, left bundle branch block, second- or third-degree heart block)
  2. Patients with a mean of two sitting systolic blood pressure (SBP) readings equal to or greater than 160 mm Hg or sitting diastolic blood pressure (DBP) equal to or greater than 100 mm Hg at Visits 1 (Screening) and 2 (Baseline/Randomization) using an automatic office blood pressure monitor
  3. Patients with pacemakers
  4. Patients with an upper arm circumference less than 24 cm or greater than 42 cm in their nondominant arm
  5. Patients with evidence of active liver disease (levels of aspartate aminotransferase, alanine aminotransferase, and/or alkaline phosphatase > 1.5× the upper limit of the normal range for the clinical laboratory performing the test)
  6. Patients with renal impairment (estimated creatinine clearance < 50 mL/min)
  7. Patients with documented autoimmune disease. Patients diagnosed with Hashimoto or Grave disease that has been stable for 3 months prior to Visit 1 (Screening) will be allowed to enroll
  8. Patients with current systemic infection (eg, human immunodeficiency virus, hepatitis)
  9. Patients with active cancer, except basal cell carcinoma. Patients taking prophylactic tamoxifen (or other antiestrogen agents) because of a family history of breast cancer or patients taking tamoxifen (or other antiestrogen agents) but who are at least 1 year post-active treatment of breast cancer, may be enrolled
  10. Patients with a current life expectancy of less than 1 year
  11. Patients with active peptic ulcer disease or history of inflammatory bowel disease or celiac sprue
  12. Patients with pulmonary dysfunction or severe chronic obstructive pulmonary disease that, in the Investigator's judgment, could interfere with study participation and completion
  13. Patients with unstable endocrine disease, including unstable diabetes or thyroid disease. Disorders that have been stable for the preceding 3 months will be acceptable
  14. Male patients with prostatic enlargement or other genitourinary disorders who might be at significant risk for dysuria and/or urinary retention while taking agents with noradrenaline-reuptake inhibition properties
  15. Pregnant or breastfeeding patients
  16. Any other conditions (such as epilepsy) that, in the Investigator's judgment, would indicate that the patient is unsuitable for the study (eg, might interfere with study conduct, confound the interpretation of study results, endanger the patient)
* Treatment-Related Criteria

  1. Patients who have received treatment with an experimental agent within the last 30 days prior to Visit 1 (Screening). Patients who have completed previous milnacipran studies (ie, all respective protocol-related study procedures have been completed by the patient) are eligible to participate. Any patients who failed screening in previous milnacipran studies may be re-evaluated, and eligible patients may enroll. Patients currently enrolled in Study MLN-MD-06 are not eligible to participate
  2. Patients who are receiving concomitant therapy with digitalis (digoxin) preparations. (Note: Patients should not undergo washout of digoxin; therefore, patients on digoxin should not be enrolled in the study)
  3. Patients who are receiving concomitant therapy with monoamine oxidase inhibitors, tricyclics, tetracyclics, SSRIs, noradrenaline or noradrenaline-serotonin (NSRI) reuptake inhibitors, SNRIs, St. John's Wort, and/or other agents marketed as antidepressants and are unable to washout or for whom washout is inadvisable*
  4. Patients who are receiving concomitant therapy with pregabalin (Lyrica) or gabapentin (Neurontin) and are unable to washout or for whom washout is inadvisable*
  5. Patients who are receiving concomitant therapy with stimulant medications such as those used to treat attention deficit disorder/attention deficit hyperactivity disorder (eg, amphetamine/dextroamphetamine [Adderall], methylphenidate, dextroamphetamine) or the fatigue associated with sleep apnea or shift work (eg, modafinil) and are unable to washout or for whom washout is inadvisable*
  6. Patients who are receiving concomitant therapy with anorectic agents such as diethylpropion , sibutramine (Meridia), and phentermine (Adipex) and are unable to washout or for whom washout is inadvisable*
  7. Patients who require the use of agents affecting serotonin pharmacology, such as ondansetron (Zofran), granisetron (Kytril), and/or dolasetron (Anzemet)
  8. Patients who require doses of guaifenesin greater than 2400 mg/d (approximately 24 teaspoons)
* Occupational Criteria

  1. Patients whose occupation requires them to work nocturnal hours (eg, 11 PM to 7 AM)
* ABPM Criteria

  1. Patients whose ABPM results at Visit 2 (Baseline/Randomization) do not satisfy ABPM inclusion/exclusion criteria outlined in the ABPM training manual

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allan Spera, Study Director — Forest Laboratories
Locations (38):
- United States (38):
  - Site #032, Birmingham, Alabama
  - Site #035, Birmingham, Alabama
  - Site #038, Phoenix, Arizona
  - Site #019, Pismo Beach, California
  - Site #016, San Diego, California
  - Site #008, Walnut Creek, California
  - Site #037, Delray Beach, Florida
  - Site #025, Jacksonville, Florida
  - Site #009, Ocala, Florida
  - Site #011, Orlando, Florida
  - Site #036, Tampa, Florida
  - Site #006, Atlanta, Georgia
  - Site #030, Libertyville, Illinois
  - Site #018, Evansville, Indiana
  - Site #034, Indianapolis, Indiana
  - Site #004, Worchester, Massachusetts
  - Site #013, Springfield, Missouri
  - Site #021, Albuquerque, New Mexico
  - Site #005, East Syracuse, New York
  - Site #010, Rochester, New York
  - Site #029, Charlotte, North Carolina
  - Site #022, Winston-Salem, North Carolina
  - Site #002, Cleveland, Ohio
  - Site #017, Toledo, Ohio
  - Site #023, Eugene, Oregon
  - Site #007, Eugene, Oregon
  - Site #001, Medford, Oregon
  - Site #026, Mechanicsburg, Pennsylvania
  - Site #014, Greer, South Carolina
  - Site #027, Bristol, Tennessee
  - Site #024, Memphis, Tennessee
  - Site #031, Nashville, Tennessee
  - Site #028, Sugarland, Texas
  - Site #003, Salt Lake City, Utah
  - Site #012, Woodstock, Vermont
  - Site #020, Richmond, Virginia
  - Site #015, Bellingham, Washington
  - Site #033, Racine, Wisconsin

REFERENCES:
- [Derived] Trugman JM, Palmer RH, Ma Y. Milnacipran effects on 24-hour ambulatory blood pressure and heart rate in fibromyalgia patients: a randomized, placebo-controlled, dose-escalation study. Curr Med Res Opin. 2014 Apr;30(4):589-97. doi: 10.1185/03007995.2013.861812. Epub 2013 Nov 20. PMID 24188161

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was from October 15, 2007 to April 16, 2008 at 38 centers in the US.
Pre-assignment Details: Following 1-to-4 week washout/single-blind placebo lead-in period, patients were randomized (2:1) to one of the treatment groups, milnacipran or placebo, respectively; and orally treated with study medication for 7-week, double-blind treatment period (Visit 2 to 6), followed by a 2-week single-blind placebo discontinuation period (Visit 6 to 8).
Groups:
- Placebo: ITT N= 93, OC analyzed n=89
- Milnacipran: Milnacipran 100 to 200 mg/day tablet, oral administration, BID.
Period: Overall Study
Arm/Group | Placebo | Milnacipran
Started | 111 | 210
Completed | 86 | 160
Not Completed | 25 | 50
Not completed — Adverse Event | 10 | 34
Not completed — Lack of Efficacy | 2 | 1
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Lost to Follow-up | 4 | 5
Not completed — Protocol Violation | 2 | 2
Not completed — did not meet criteria, non-compliance | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Milnacipran | Total
Number analyzed (Participants) | 111 | 210 | 321
Age Continuous [Mean (Standard Deviation); unit: years] | 48.9 (11.1) | 48.3 (10.9) | 48.5 (11.0)
Age, Customized [Number; unit: participants]
  < 20 years | 1 | 2 | 3
  20-59 years | 91 | 174 | 265
  >= 60 years | 19 | 34 | 53
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 198 | 307
  Male | 2 | 12 | 14
Region of Enrollment [Number; unit: participants]
  United States | 111 | 210 | 321

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Systolic Blood Pressure Following 12-hour Period Post-AM Dose at Visit 4
Description: Change from baseline to Visit 4 in mean systolic blood pressure (SBP) based on ambulatory blood pressure monitor (ABPM) is defined as the mean SBP value at Visit 4 minus the corresponding mean SBP value at baseline in the same 12-hour period post-AM dose.
Time Frame: 4 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: Normotensive: ITT N=42, OC analyzed n=39; hypertensive: ITT N=51, OC analyzed n=50
- Milnacipran: Normotensive: ITT N=93, OC analyzed n=92; hypertensive: ITT N=88, OC analyzed n=84
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 89 | 176
mm Hg
  Change in SBP in Normotensive Patients | -0.9 (1.0) | 4.0 (0.8)
  Change in SBP in Hypertensive Patients | 0.2 (1.1) | 3.7 (1.0)

2. Secondary Outcome: Change From Baseline in Mean Systolic Blood Pressure /Diastolic Blood Pressure for 12-hour Period Post-AM Dose at Visit 4
Description: Change from baseline to Visit 4 in mean SBP/DBP based on ABPM is defined as the mean SBP/DBP values at Visit 4 minus the corresponding mean SBP/DBP values at baseline in the same 12-hour period post-AM dose.
Time Frame: 4 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Milnacipran: ITT N= 181, OC analyzed n=176
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 89 | 176
mm Hg
  Change in Systolic Blood Pressure | -0.3 (0.8) | 3.8 (0.6)
  Change in Diastolic Blood Pressure | -0.3 (0.6) | 4.2 (0.5)

3. Primary Outcome: Change From Baseline in Mean Systolic Blood Pressure Following 12-hour Period Post-AM Dose at Visit 6
Description: Change from baseline to Visit 6 in mean systolic blood pressure based on ABPM is defined as the mean SBP value at Visit 6 minus the corresponding mean SBP value at baseline in the same 12-hour period post-AM dose.
Time Frame: 7 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d, followed by 1 week at 150 mg/d and 2 weeks of 200 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: Normotensive: ITT N= 42, OC analyzed n=37; hypertensive: ITT N=51, OC analyzed n=47
- Milnacipran: Normotensive: ITT N= 93, OC analyzed n=82; hypertensive: ITT N=88, OC analyzed n=80
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 84 | 162
mm Hg
  Change in SBP in Normotensive Patients | 0.1 (1.3) | 5.5 (0.9)
  Change in SBP in Hypertensive Patients | -0.9 (1.4) | 4.4 (1.0)

4. Secondary Outcome: Change From Baseline in Mean SBP/DBP Following 12-hour Period Post-AM Dose at Visit 6
Description: Change from baseline to Visit 6 in mean SBP/DBP based on ABPM is defined as the mean SBP/DBP value at Visit 6 minus the corresponding mean SBP/DBP value at baseline in the same 12-hour period post-AM dose.
Time Frame: 7 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d, followed by 1 week at 150 mg/d and 2 weeks of 200 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach.
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Placebo: ITT N=93, OC analyzed n=84
- Milnacipran: ITT N=181, OC analyzed n=162
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 84 | 162
mm Hg
  Change in Systolic Blood Pressure | -0.4 (1.0) | 5.0 (0.7)
  Change in Diastolic Blood Pressure | -0.5 (0.7) | 5.0 (0.5)

5. Secondary Outcome: Change From Baseline in Mean Heart Rate (HR) Following 24-hour Treatment at Visit 4
Description: Change from baseline to Visit 4 in HR based on ABPM is defined as the mean HR value at Visit 4 minus the corresponding mean HR value at baseline in the same 24-hour period.
Time Frame: 4 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach.
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 89 | 176
bpm
  Change in Heart Rate | -1.0 (0.6) | 11.7 (0.5)

6. Secondary Outcome: Change From Baseline in Mean HR Following 24-hour Treatment at Visit 6
Description: Change from baseline to Visit 6 in HR based on ABPM is defined as the mean HR value at Visit 6 minus the corresponding mean HR value at baseline in the same 24-hour period.
Time Frame: 7 weeks (1 week of dose-escalation, 3 weeks of 100 mg/d, followed by 1 week at 150 mg/d and 2 weeks of 200 mg/d)
Population: The analysis was based on Intent-To-Treat (ITT) population using Observed Cases (OC) approach.
Measure: Mean (Standard Error); unit: bpm
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 84 | 162
bpm
  Change in Heart Rate | -1.6 (0.7) | 12.9 (0.6)

ADVERSE EVENTS:
Time Frame: 7 weeks double-blind treatment period followed by 2 weeks single-blind placebo discontinuation period.
Description: For SAEs, 3 of 210 affected in double-blind treatment period & 3 of 164 affected in single-blind placebo discontinuation period in milnacipran arm; 1 of 111 affected in double-blind treatment period & 0 of 88 affected in single-blind placebo discontinuation period in placebo arm.
Arm/Group | Placebo | Milnacipran
Serious Adverse Events (participants affected / at risk) | 1/111 | 6/210
Other Adverse Events (participants affected / at risk) | 42/111 | 117/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=111) | Milnacipran (N=210)
Atrial Flutter (Cardiac disorders) | 0 | 1
Hypertensive Crisis (Vascular disorders) | 0 | 1
Uterine Haemorrhage (Reproductive system and breast disorders) | 0 | 1
Complicated Migraine (Nervous system disorders) | 1 | 0
Chest Pain (General disorders) | 0/88 | 1/164
Coronary Artery Stenosis (Cardiac disorders) | 0/88 | 1/164
Diarrhoea (Gastrointestinal disorders) | 0/88 | 1/164
Hiatus Hernia (Gastrointestinal disorders) | 0/88 | 1/164
Multiple Injuries (Injury, poisoning and procedural complications) | 0/88 | 1/164
Non-Cardiac Chest Pain (General disorders) | 0/88 | 1/164
Pericardial Effusion (Cardiac disorders) | 0/88 | 1/164
Periorbital Cellulitis (Infections and infestations) | 0/88 | 1/164
Peritoneal Haemorrhage (Gastrointestinal disorders) | 0/88 | 1/164
Rib Fracture (Injury, poisoning and procedural complications) | 0/88 | 1/164
Road traffic accident (Injury, poisoning and procedural complications) | 0/88 | 1/164
Sinusitis (Infections and infestations) | 0/88 | 1/164
Spelnic Rupture (Injury, poisoning and procedural complications) | 0/88 | 1/164
Vomiting (Gastrointestinal disorders) | 0/88 | 1/164
Wrist Fracture (Injury, poisoning and procedural complications) | 0/88 | 1/164
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Milnacipran (N=210)
Nausea (Gastrointestinal disorders) | 11 | 48
Headache (Nervous system disorders) | 5 | 28
Constipation (Gastrointestinal disorders) | 1 | 23
Tachycardia (Cardiac disorders) | 1 | 20
Dizziness (Nervous system disorders) | 2 | 16
Vomiting (Gastrointestinal disorders) | 2 | 16
Palpitations (Cardiac disorders) | 3 | 14
Hot Flush (Vascular disorders) | 2 | 13
Insomnia (Psychiatric disorders) | 9 | 12
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 8
Urinary Tract Infection (Infections and infestations) | 7 | 7
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 6 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release & can embargo communications re: results for 90 days from time submitted to sponsor for review. PI shall not disclose sponsor's confidential info. Upon sponsor's request, PI shall delete any proprietary info & shall not include raw data in pub. On sponsor's request, PI shall delay submission for any pub while sponsor files patent apps. If trial is multi-center, PI agrees that first publication shall be a multi-center pub.